CLINICAL TRIAL: NCT01436136
Title: Effectiveness of Team Intervention Over 12 Months in Reducing Modifiable CVD Risk Factors on Framingham 10yr Risk Scores Outcomes in HIV-1 Subjects on Antiretroviral Therapy
Brief Title: Reducing Cardiovascular Disease (CVD) Risk in HIV on Antiretroviral Therapy Over 12 Months
Acronym: CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holdsworth House Medical Practice (Other)
Responsible Party: Principal Investigator, Dr. Mark Bloch, Doctor, Holdsworth House Medical Practice
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Reducing CVD risk in HIV
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: HIV-1 Infection; Cardiovascular Disease
Keywords: Cardiovascular disease; HIV; Antiretroviral treatment; team interventions; Framingham risk score
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Patients randomised to the intervention group will follow an intensive 52 week period using a clinical protocol aimed to manage CVD risk in HIV individuals with the use of regular visits to a nurse led CVD risk management clinic, within a multi disciplinary approach to care with the involvement of treating physicians, nurses, dieticians, smoking cessation advisors and an exercise physiologist or personal trainer with the aim to reach their individualised CVD risk target.
  Interventions: Other: Control
- Usual care (control) group (Active Comparator): Within the context of an open, cohort study, GPs managing matched control patients allocated usual care will be unaware of the details of the intervention arm and asked to apply their usual pattern of patient visits and treatment strategies to achieve optimal reduction of CVD risk.
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Control — GPs managing matched control patients allocated usual care will be unaware of the details of the intervention arm and asked to apply their usual pattern of patient visits and treatment strategies to achieve optimal reduction of CVD risk.
  Arms: Intervention group
Other: Intervention Group — Patients randomised to the intervention group will follow an intensive 52 week period using a clinical protocol aimed to manage CVD risk in HIV individuals with the use of regular visits to a nurse led CVD risk management clinic, within a multi disciplinary approach to care with the involvement of treating physicians, nurses, dieticians, smoking cessation advisors and an exercise physiologist or personal trainer with the aim to reach their individualised CVD risk target.
  Arms: Usual care (control) group

SUMMARY:
This is a cohort study which follows two groups of participants over a 12 months period. One group will access a team approach to care with the aim of reducing their cardiovascular disease (CVD) risks from a team of doctors, nurses and health care professionals. The other group will continue to access standard care from their treating doctor. Both groups will have CVD risk score evaluated after a 12 month period.

The team care approach will involve specific tests to measure CVD risk as well as smoking cessation, exercise and dietary advice and support, including monitoring such as blood pressure and cholesterol levels

ELIGIBILITY:
intervention study intervention arm

Inclusion criteria:

1. Documented HIV-1 infection
2. Age 50 years or older
3. Stable on ART ≥ 3/12
4. Undetectable plasma HIV RNA (< 50 copies/ml)
5. Moderate or high Framingham CVD risk score
6. Life expectancy > 12 months
7. Regular patient under care of non-director physician
8. Willing to adhere to pharmacological CVD risk reduction intervention
9. Willing to participate in lifestyle change advice intervention

Exclusion criteria for intervention study

1. Life expectancy < 1yr
2. Unable to undertake exercise
3. Drug dependency
4. Cognitive impairment affecting ability to participate in study
5. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5mI U/ml)
6. Women of childbearing potential who are unwilling to use reliable contraception for the duration of the study

Inclusion criteria for intervention study control arm (Group 2)

1. Documented HIV-1 infection
2. Age 50 years or older
3. Stable on ART ≥3/12
4. Undetectable plasma HIV RNA (<50 copies/ml)
5. Moderate or high Framingham risk score (>10%)
6. Life expectancy > 12 months
7. Regular patient under care of non-director physician

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is percentage of patients with a reduction of Framingham risk score of at least 10% at week 52. | 12 months
  The primary outcome measure is percentage of patients with a reduction of Framingham risk score of at least 10% at week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Bloch, Principal Investigator — Australian Health Practitioner Regulation Agency
Locations (1):
- Holdsworth House Medical Practice, Sydney, New South Wales, Australia